CLINICAL TRIAL: NCT05731687
Title: Bifurcation PCI With a Hybrid Strategy With Drug Eluting Balloons Versus a Stepwise Provisional Two-stent Strategy. A Randomized Controlled Trial and Registry
Brief Title: Bifurcation PCI With a Hybrid Strategy With Drug Eluting Balloons Versus a Stepwise Provisional Two-stent Strategy
Acronym: Hybrid DEB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cathreine BV (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other); Albert Schweitzer Hospital (Other); Onze Lieve Vrouwe Gasthuis (Other); Maasstad Hospital (Other); The Elisabeth-TweeSteden Hospital (Other); St. Antonius Hospital (Other); Frisius Medisch Centrum (Other); Meander Medical Center (Other); VieCuri Medical Centre (Other); Haga Hospital (Other); Rijnstate Hospital (Other); Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, Koen Teeuwen, Koen Teeuwen, MD, PhD, Principal Investigator, Cathreine BV
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21112022
Record Dates: First submitted 2023-01-25; First posted 2023-02-16 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Coronary Bifurcation Lesion
Keywords: Coronary bifurcation lesion; Coronary artery disease; Drug-eluting balloon; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to either hybrid DEB approach or two-stent strategy
Who Masked: Participant
Masking Description: This is a single-blinded study. The patients are blinded for the allocated therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid DEB (Other): Patients randomized to hybrid DEB group will receive application of DEB in the side branch.
  Interventions: Other: Hybrid DEB approach with drug-eluting balloon
- Two-stent strategy (Other): Patients randomized to two-stent strategy will receive implantation of a second DES in the side branch, using Culotte or TAP/T technique.
  Interventions: Other: Two-stent strategy

INTERVENTIONS:
Other: Hybrid DEB approach with drug-eluting balloon — If a patient is randomized to the hybrid DEB approach, lesion preparation of the SB with non-compliant balloon (NC) is mandatory before DEB application. The application of DEB can be performed if acceptable result of the lesion preparation is obtained (at least TIMI III flow and no flow limiting dissection). The drug- eluting balloon used in this study is the CE- marked Magic Touch Sirolimus Coated Balloon Catheter (Concept Medical, Gujarat, India). The size of the DEB is measured on a ratio 1:1 on reference diameter of the SB. The DEB balloon is inflated for 60 seconds, or two times more than 30 seconds if long duration inflations are not possible. Finally low pressure kissing inflation with the same DEB in place, and Proximal Optimization Therapy (POT) are performed. In case of SB occlusion, or flow limiting dissections in non-Left Main (LM) bifurcations and < TIMI 3 flow or 70-99% residual stenosis in LM bifurcations, cross- over to two-stent technique is performed.
  Arms: Hybrid DEB
Other: Two-stent strategy — When randomized to the conventional two-stent strategy, TAP/T or Culotte stenting is performed. First lesion preparation of the SB is mandatory. The drug-eluting stent (Supraflex stent) can be placed in the SB if acceptable result of the lesion preparation is obtained and is measured on a 1:1 ratio on reference diameter of the SB. Finally, kissing inflation and POT are mandatory.
  Arms: Two-stent strategy

SUMMARY:
The optimal treatment of coronary bifurcation lesions is complex and remains subject of current research. There is ongoing debate about the optimal strategy for bifurcations with upfront two-stent strategy or provisional one-stent strategy. Current European Society of Cardiology (ESC) guidelines advise a provisional approach with optional stepwise two-stent strategy in case of suboptimal result of the side branch (SB). However, a two-stent strategy (either upfront and stepwise) caries technical difficulties and is associated with increased procedure duration and costs and higher exposure of the patient to radiation and contrast. Therefore there is upcoming interest in the use of a drug-eluting balloon (DEB) in the side branch of bifurcation lesions after provisional approach. Drug-eluting balloons are conventional semi-compliant angioplasty balloons covered with an anti-proliferating drug, which is released into the vessel wall during inflation.

Several small pilot studies have successfully investigated a hybrid approach with use of DEB in addition to the provisional strategy. This hybrid approach has shown to be safe and feasible, however no large trials have been performed comparing this with current two-stent bifurcation strategies.

The aim of this randomized controlled, single blinded, multicenter trial is to investigate whether a hybrid DEB approach is non-inferior to a stepwise provisional two-stent strategy in patients with de novo bifurcation lesions and a suboptimal result of the SB after provisional approach.

Patients included in this study will receive PCI using provisional approach (implantation of drug-eluting stent (DES) in the main branch). Patients with an unsatisfactory result of the SB after provisional PCI (≥ 70% residual stenosis and/or diminished flow < Thrombolysis in Myocardial Infarction (TIMI) III) will be randomized in a 1:1 ratio to receive the Hybrid DEB approach or the two-stent strategy. Patients with a satisfactory result of the side branch after provisional PCI will be included in a registry.

Follow-up will be performed at 12 months and at the anticipated median 2 year follow-up with a minimum follow-up of 1 year in each subject by either a phone call or outpatient clinic visit. During follow-up information regarding cardiovascular drug use, hospitalizations, invasive and non-invasive diagnostic tests, angina status and SAE's is obtained.

ELIGIBILITY:
Inclusion Criteria:

* Significant de novo bifurcation lesion (main vessel and side branch diameter ≥ 2.5mm, diameter stenosis of the main vessel ≥ 70% and of the side branch ≥ 50% or in intermediate stenosis FFR ≤ 0.80 or iFR ≤ 0.89)
* Stable coronary artery disease or stabilized acute coronary syndrome
* Age ≥ 18 years
* Acceptable candidate for treatment with a drug eluting stent

Exclusion Criteria:

* Unstable clinical condition
* Previous PCI with stent implantation in the target lesion(s)
* Known comorbidity with a life expectancy of <2 year
* Active bleeding requiring medical attentions (BARC >2 at index PCI)
* Pregnancy
* Unable to provide consent for any other reason
* Participation in another stent or drug trial
* Known hypersensitivity or allergy for asprin, clopidogrel, ticagrelor, prasugrel, cobalt chromium, sirolimus, to excipients with phospholipid or related origins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death, periprocedural or spontaneous myocardial infarction (MI) and/or target vessel revascularization (TVR) | Anticipated median 2 year follow-up after the date of randomization, with a minimum follow-up in all subjects of 1 year
  Composite of all-cause death, periprocedural (according to the SCAI/ARC II definition and a secondary analysis according to the 4th universal definition) or spontaneous (according to the 4th universal definition) myocardial infarction (MI) and/or target vessel revascularization (TVR) at the anticipated median 2 year

SECONDARY OUTCOMES:
Procedural success | Discharge, 12 months and the anticipated median 2 year follow-up after the date of randomization
  Procedural success defined as successful stent delivery with final core lab (defined as TIMI flow of III, angiographic in-stent MB and SB diameter stenosis ≤30%, or ≤50% after DEB in the side branch) and absence of in-hospital major adverse cardiac and cerebrovascular events (MACCE, defined as all cause death, spontaneous MI, TVR, stoke) at discharge, 12 months and the anticipated median 2 year
Target vessel failure (TVF) | Discharge, 12 months and the anticipated median 2 year follow-up after the date of randomization
  Target vessel failure (TVF), defined as cardiac death, target vessel spontaneous MI, TVR at discharge, 12 months and the anticipated median 2 year
Major adverse cardiac events (MACE) | Discharge, 12 months and the anticipated median 2 year follow-up after the date of randomization
  Major adverse cardiac events (MACE), defined as all-cause death, spontaneous MI, repeat revascularization at discharge, 12 months and the anticipated median 2 year
Individual components of MACE and TVF | Discharge, 12 months and the anticipated median 2 year follow-up after the date of randomization
  Individual components of MACE and TVF (All-cause death, cardiac death, periprocedural of spontaneous MI, target vessel revascularization, target vessel spontaneous MI) at discharge, 12 months and the anticipated median 2 year
Periprocedural MI | 48 hours after the Percutaneous Coronary Intervention (PCI)
  Periprocedural MI within 48 hours after procedure, according to the SCAI/ARC II definition, secondary analysis according to the 4th universal definition
Major intraprocedural complications | The end of the PCI
  Major intraprocedural complications, defined as type C-F dissections, perforations, slow flow or no reflow (< TIMI III), thrombus, major side branch occlusion (>2mm) during the index procedure
Probable and definite stent thrombosis | Discharge, 12 months and the anticipated median 2 year follow-up after the date of randomization
  Probable and definite stent thrombosis, defined as Angiographic confirmation of stent thrombosis, or any myocardial infarction that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause at discharge, 12 months and the anticipated median 2 year
Major bleeding, defined as BARC type 2-5 | Discharge after the PCI
  Major bleeding, defined as BARC type 2-5 at discharge
Contrast volume used during the PCI procedure | The end of the PCI
  Contrast volume used during the PCI procedure (in ml)
Radiation exposure of the patient, measured in DAP and AirKerma | The end of the PCI
  Radiation exposure of the patient, measured in DAP and AirKerma during the PCI procedure
Procedural time, measured in minutes, defined as time from first to last procedural angiography image | The end of the PCI
  Procedural time, measured in minutes, defined as time from first to last procedural angiography image
Total procedural costs (in euro's) per patient stratified to treatment group | The end of the PCI
  Total procedural costs (in euro's) per patient stratified to treatment group
Percentage of stent expansion in proximal and distal main branch and side branch, measured with intracoronary imaging (OCT or IVUS) | The end of the PCI
  Percentage of stent expansion in proximal and distal main branch and side branch, measured with intracoronary imaging (OCT or IVUS)
Final minimal lumen and stent area post stenting in the proximal and distal main branch measured with intracoronary imaging (OCT or IVUS) | The end of the PCI
  Final minimal lumen and stent area post stenting in the proximal and distal main branch measured with intracoronary imaging (OCT or IVUS)
Dissections in the proximal and distal main branch and side branch, measured using intracoronary imaging (OCT or IVUS) | The end of the PCI
  Dissections in the proximal and distal main branch and side branch, measured using intracoronary imaging (OCT or IVUS)
Core Lab Assessed initial TIMI flow main branch and side branch | During the Coronary Angiography (CAG), before the PCI
  Core Lab Assessed initial TIMI flow main branch and side branch
Core Lab Assessed Lesion Length (in mm) | During the CAG, before the PCI
  Core Lab Assessed Lesion Length (in mm)
Core Lab Assessed percentage diameter stenosis main branch and side branch | During the CAG, before the PCI
  Core Lab Assessed percentage diameter stenosis main branch and side branch
Core Lab Assessed reference diameter (in mm) proximal main branch and side branch | During the CAG, before the PCI
  Core Lab Assessed reference diameter (in mm) proximal main branch and side branch
Core Lab Assessed minimal lumen diameter (in mm) main branch and side branch | During the CAG, before the PCI
  Core Lab Assessed minimal lumen diameter (in mm) main branch and side branch
The severity of calcification main branch and side branch, Core Lab Assessed | During the CAG, before the PCI
  The severity of calcification main branch and side branch, Core Lab Assessed
Core Lab Assessed Bifurcation angle | During the CAG, before the PCI
  Core Lab Assessed Bifurcation angle
Core Lab Assessed syntax I score as absolute value | During the CAG, before the PCI
  Core Lab Assessed syntax I score as absolute value
Bifurcation medina score | During the CAG, before the PCI
  Bifurcation medina score
Core Lab Assessed final TIMI flow main branch and side branch | The end of the PCI
  Core Lab Assessed final TIMI flow main branch and side branch
Core Lab Assessed residual dissection (type A-F) after PCI in the main branch and/or side branch | The end of the PCI
  Core Lab Assessed residual dissection (type A-F) after PCI in the main branch and/or side branch
Core Lab Assessed residual in-stent and in-segment stenosis (in %) after PCI | The end of the PCI
  Core Lab Assessed residual in-stent and in-segment stenosis (in %) after PCI
Core Lab Assessed minimal lumen diameter (in mm) main branch and side branch post PCI | The end of the PCI
  Core Lab Assessed minimal lumen diameter (in mm) main branch and side branch post PCI
Core Lab Assessed percentage diameter stenosis main branch and side branch post PCI | The end of the PCI
  Core Lab Assessed percentage diameter stenosis main branch and side branch post PCI
Core Lab Assessed acute lumen gain (in mm) main of the branch and side branch after PCI | The end of the PCI
  Core Lab Assessed acute lumen gain (in mm) main of the branch and side branch after PCI
Core Lab Assessed Procedural coronary thrombus | The end of the PCI
  Core Lab Assessed Procedural coronary thrombus, defined as yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dillen DMM, Vlaar PJ, Vermeer AJE, Paradies V, van Kuijk JP, Vink MA, Oemrawsingh RM, Hofma SH, Magro M, Remkes WS, de Smet BJGL, van Rees JB, Somi S, Halim J, Zimmermann FM, Wijnbergen IF, Tijssen JGP, Tonino PAL, Teeuwen K. Bifurcation PCI with a hybrid strategy with drug- eluting balloons versus a stepwise provisional two- stent strategy: Rationale and design of the hybrid DEB study. Am Heart J. 2023 Dec;266:168-175. doi: 10.1016/j.ahj.2023.09.010. Epub 2023 Oct 6. PMID 37806333